CLINICAL TRIAL: NCT03725670
Title: Direct Lentiviral TYF-ARSA Injection Gene Therapy for Metachromatic Leukodystrophy (MLD)
Brief Title: Direct Lentiviral Injection Gene Therapy for MLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-18005
Record Dates: First submitted 2018-09-25; First posted 2018-10-31 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Metachromatic Leukodystrophy (MLD)
Keywords: Metachromatic leukodystrophy (MLD); lentiviral vector; Intrathecal injection; Intravenous injection
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lentivirus-mediated delivery of ARSA to the CNS and the body (Experimental): Intrathecal and intravenous injections with lentiviral TYF-ARSA vector carrying the functional gene
  Interventions: Genetic: Intrathecal and intravenous LV gene therapy

INTERVENTIONS:
Genetic: Intrathecal and intravenous LV gene therapy — Direct IT and IV LV gene therapy to deliver high levels of LVs at 1-2×10^9 transduction units/ml which carry a normal ARSA gene

SUMMARY:
This is a Phase I/II clinical trial of gene therapy for treating Metachromatic leukodystrophy (MLD) using a safety and efficacy improved self-inactivating lentiviral vector TYF-ARSA to functionally correct the genetic defect. The primary objectives are to evaluate the safety and efficacy of the direct gene transfer clinical protocol.

DETAILED DESCRIPTION:
Metachromatic leukodystrophy (MLD) is a rare lysosomal storage disease. This disease is an inherited single gene autosomal recessive defect. MLD is caused by a mutation in the ARSA gene encoding arylsulfatase A which leads to a deficiency in sulfatide degradation, resulting in its accumulation in oligodendrocytes, Schwann cells and neurons. A critical level of sulfatide storage can trigger demyelination, the hallmark of MLD, which results in multiple neurological symptoms. MLD has different onset ages including late infancy (1-2 years), adolescence (4 years-before sexual maturity) and adulthood (after sexual maturity). MLD patients are normally rescued by hematopoietic stem cell transplantation (HSCT) from a matched healthy donor. However, HSCT must be performed at a very early stage of the disease thus restricting its therapeutic opportunies in MLD patients. This trial aims to treat MLD using a safety and efficacy improved self-inactivating lentiviral vector (LV) carrying a functional MLD gene to correct the genetic defect by intrathecal (IT) and intravenous (IV) injections to delivery the lentiviral vector carrying a normal ARSA gene to correct the genetic defect. The primary objectives are to evaluate the safety of the improved LV TYF-ARSA and the direct injection gene transfer clinical protocol, the efficacy of degradative metabolite in patients after treatment, vector integration profile, and finally the long-term correction of the related pathological symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. MLD patient age >= 1 month
2. ARSA gene sequence analysis to confirm MLD mutations
3. Scoring system for brain MR Imaging confirmed MLD
4. Parent / guardian / patient signing informed consent
5. Patients and their families have a strong willingness to participate in clinical trials, and are willing to bear all the consequences caused by the failure of the trial, and sign an informed consent form

Exclusion Criteria:

1. HIV positive patients
2. Patients who are experiencing uncontrolled viral, bacterial or fungal infections, malignant tumors, heart abnormalities, liver dysfunction, or renal insufficiency
3. Cannot perform an MRI
4. Infection or dermatosis at pre-injection site
5. Any condition that may increase the subjects' risk or interfere with the results of the trial. In addition to MLD, there are other neurological disorders.

Ages: 1 Month to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of IT and IV injections of lentiviral TYF-ARSA | up to 1 year follow up
  Safety of IT and IV injections of lentiviral TYF-ARSA, determined by number of participants with treatment-related adverse events (AEs), according to scheduled assessments, vital signs, & physical examinations as assessed by CTCAE v4.0. AEs & clinically significant abnormalities (meeting grade 3, 4, or 5 criteria according to CTCAE) will be summarized by maximum intensity & relationship to the study drug(s). The grade of AEs will be summarized if related to the treatment.
Altered disease progression | up to 3 year follow up after treatment
  Altered disease progression based on biochemical analysis.
Altered disease progression | up to 3 year follow up after treatment
  Altered disease progression based on MRI brain imaging analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Ph.D, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Lung-Ji Chang, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No